CLINICAL TRIAL: NCT03143920
Title: Hyperbaric Oxygen Therapy for Inflammatory Conditions of the Urinary Bladder: A Feasibility Trial
Brief Title: Hyperbaric Oxygen Therapy for Inflammatory Conditions of the Urinary Bladder
Acronym: HBOTCICrUTI
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No funding to continue
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Ian Grover, MD, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBOTurology.2017
Record Dates: First submitted 2017-05-02; First posted 2017-05-08 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Chronic Interstitial Cystitis; Painful Bladder Syndrome; Recurrent Urinary Tract Infection
Keywords: hyperbaric oxygen; inflammation; chronic disease; urinary bladder; urinary tract infection; recurrent urinary tract infection; painful bladder syndrome; chronic pain; hypoxia; bacterial infection
MeSH Terms: conditions — Cystitis, Interstitial; Urinary Tract Infections; Inflammation; Chronic Disease; Chronic Pain; Hypoxia; Bacterial Infections | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Prospective pilot study to test feasibility of treating patients with chronic inflammatory conditions of the urinary bladder with hyperbaric oxygen therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Hyperbaric Oxygen (Experimental): Hyperbaric oxygen therapy-2.4 atmosphere absolute for 90 minutes with 2-five minute air breaks administered daily, 5 days per week for 8 weeks total treatment.
  Interventions: Combination Product: Hyperbaric Oxygen Therapy-

INTERVENTIONS:
Combination Product: Hyperbaric Oxygen Therapy- — Hyperbaric oxygen therapy provides 100% medical grade oxygen at 2.4 atmospheres of absolute pressure with a Class A multiple person chamber or Class B single person chamber. Hyperbaric chambers are classified as a Class II medical device and have been FDA cleared.

SUMMARY:
Pilot study to determine feasibility for treating patients with two chronic inflammatory conditions of the urinary bladder: chronic interstitial cystitis and recurrent urinary tract infections using a standardized hyperbaric oxygen treatment plan. Presently there are no good treatments for these conditions and hyperbaric oxygen may be a safe and readily accessible therapy as it has proven successful an another type of chronic inflammatory condition of the urinary bladder known as "radiation cystitis". The study will determine if patients will consider this an acceptable treatment for their conditions and that it is well tolerated.

DETAILED DESCRIPTION:
The primary object is to determine the feasibility of treating patients diagnosed with either CIC/PBS or rUTI with daily hyperbaric oxygen for a total of 40 treatment sessions during an 8-10 week time period. We wish to better understand the demand and degree of adherence for daily HBOT in these two patient populations to inform future planning and design of randomized, sham controlled and double-blind studies. Given the refractory nature of these two diagnoses, a secondary objective of this study is to determine if there is symptomatic improvement following HBOT compared to pretreatment symptoms using standardized patient symptomology questionnaires' (Global Response Assessment-GRA and Patient's Overall Rating of Improvement in Symptoms-PORIS questionnaires).

Patient selection will be carried out by the respective co-investigators based on standard disease definitions. CIC/PBS is defined as urinary tract pain or discomfort and dysuria that is present of > 6 months and is not due to acute urinary tract infection, stones or other pathology. These patients will be identified and recruited by Dr. C. Lowell Parsons, Co-investigator for the study. rUTI is defined as greater than 2 urinary tract infections in 6 month or greater than 3 urinary tract infections in one year. These patient will be identified and recruited by Dr. Emily Lukacz, Co-investigator. Each study will enroll 20 individuals. The study design is an observational pilot study to determine feasibility and limited efficacy. Thus the primary outcomes will be the number of patients that enroll in the study relative to the number offered enrollment and the percentage of individuals completing the prescribed 40 treatment sessions. For the secondary outcome, limited efficacy, each patient's pre-treatment clinical status will be compared to their post treatment clinical status. Thus for the CIC/PBS study both the global response assessment (GRA) and the patient's overall rating of improvement of symptoms (PORIS) will be obtained and comparison between the pre and post treatment scores will be performed. For the UTI study, the time in days to subsequent acute urinary tract infection and total number of acute UTI's during one year following completion of HBOT will be recorded and compared to that individual's prior clinical history. The dosing algorithm to be used is based on the current standard of care for the treatment of radiation cystitis for which 2.4 ATA x 90 minutes is provided daily, 5 days per week. The total duration of treatment can range from 30-60 minutes depending upon the individual patients severity of illness and response to therapy. Patients are routinely reassessed after every 10-20 treatments. Therefore we are planning to provide 2.4 ATA x 90 minutes with 2 air breaks daily, x 5 days per week x 8 weeks total for both CIC/PBS and rUTI patient population. We will allow the 40 treatments to be administered over an 8-10 week time period to provide some degree of scheduling flexibility for patients.

For this feasibility study we will determine the demand as measured by the number of patients accepting the treatment vs the total number of patients offered enrollment. We will determine the percentage successful completion of the 40 prescribed treatment sessions as the primary outcome variable. The results of the symptom questionnaires obtained at the conclusion for HBOT and by follow up telephone survey at 1, 6 and 12 months following completion of HBOT will be the secondary outcome variable. Finally, adverse events will be gathered on this patient population as per routine clinical practice. The incidence and severity of otic barotrauma, hyperoxic myopia, confinement anxiety and generalized seizures will be determined and compared to the same events experienced by the general hyperbaric patient population being treated during the same period of time.

Symptom Survey Instruments Global Response Assessment (GRA) The GRA measures overall improvement with therapy. It is now used as the primary end point in clinical trials of therapies for CIC/PBS. The assessment asks: "As compared to when you started the study [treatment], how would you rate your interstitial cystitis symptoms now?" The seven point scale is centered at zero (no change): markedly worse; moderately worse; slightly worse; no change; slightly improved; moderately improved; and markedly improved. Responders will be defined as those individuals with scores falling in the moderately and markedly improved categories.

Patient's Overall Rating of Improvement of Symptoms (PORIS) The PORIS has three questions that address the overall change in CIC/PBS, pain, and urgency after treatment as worse, no better (0% improvement), slightly improved (25%), moderately improved (50%), greatly improved (75%), or symptoms gone (100% improvement). Responders will be defined as those individuals with scores falling into the moderately or greatly improved or no symptoms categories.

ELIGIBILITY:
Inclusion Criteria:

* CIC/PBS- patients with urinary tract pain or discomfort and dysuria that is present for > 6 months and is not due to acute urinary tract infection, stones or other urinary pathology.
* rUTI- patients with greater that 2 urinary tract infections in 6 months or greater than 3 urinary tract infections in one year. A UTI is defined as - symptomatic complaints of dysuria, increased frequency of urination, and hesitancy to urinate and a clean catch urinary culture with >103 colony counts of bacteria per milliliter.

Exclusion Criteria:

* Inability to provide written informed consent
* Inability or unwillingness to adhere to 40 HBOT treatment sessions over an 8-10 week time period or to complete follow up questionnaires/telephone contacts.
* Confinement anxiety and inability to enter the hyperbaric chamber for a 90 minutes treatment session.
* Inability to effectively equalize the middle ear during changes in ambient pressure. This will include patients with a history of tympanic membrane perforation, head and neck surgery with compromised Eustachian tube function, including but not limited to tracheostomy, mastoidectomy, middle ear surgical procedures and cochlear implants.
* Presence of an indwelling urinary catheter
* Any acute or chronic urinary condition that is not rUTI or CIC/PBS- such as but not limited to urinary bladder stones, tumors, urinary retention, adynamic urinary bladder, chemotherapy related hemorrhagic cystitis, radiation cystitis or other pathology.
* Active or uncontrolled cancer diagnosis.
* Active or uncontrolled psychiatric disease.
* American Heart Association Class III or greater congestive heart failure or symptomatic coronary artery disease.
* Active or uncontrolled pulmonary diseases- including asthma, COPD, bullous lung disease, previous thoracotomy, pneumothorax or history of pneumothorax.
* Acute upper respiratory tract infection.
* End stage renal disease receiving hemo- or peritoneal dialysis
* Active or history of seizure disorder
* Hemolytic blood dyscrasias
* History of exposure to bleomycin
* Presence of a pacemaker or epidural pain pump
* Pregnant or lactating women
* Patients with type 2 diabetes
* Patients with neurovascular diseases (e.g. recent stroke)
* Patients with uncontrolled hypertension
* Patients with retinitis pigmentosa
* Patients taking the following concomitant medications: PDE5 inhibitors, carbonic anhydrase inhibitors, beta blockers, alpha blockers, nitrates.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
HBOT acceptance | Three year study period. Determination is made for this endpoint at time of initiation of HBOT
  The primary outcome will be the number of patients that enroll in the study relative to the number offered enrollment and reported as a percentage of total patients offered enrollment.
HBOT adherence | Three year study period. Determination is made for this endpoint on the date of final HBOT session.
  The number of individuals completing the prescribed 40 treatment sessions and reported as a percentage of the number of individuals who initially enrolled in the study.

SECONDARY OUTCOMES:
Pre and post treatment symptom survey for the chronic interstitial cystitis study group. | Three year study period. Determination is made for this endpoint on the date prior to first HBOT and final HBOT session and then by telephone followup at 1, 6, and 12 months following the last HBOT session.
  The global response assessment (GRA)will be obtained and comparison between the pre and post treatment scores will be performed. The GRA measures overall improvement with therapy. It is now used as the primary end point in clinical trials of therapies for CIC/PBS. The assessment asks: "As compared to when you started the study [treatment], how would you rate your interstitial cystitis symptoms now?" The seven point scale is centered at zero (no change): markedly worse; moderately worse; slightly worse; no change; slightly improved; moderately improved; and markedly improved. Responders will be defined as those individuals with scores falling in the moderately and markedly improved categories. The number of responders will be reported as a percentage of total number of individuals completing 40 HBOT sessions.
Post treatment incidence of recurrent urinary tract infection. | Three year study period. Determination of this endpoint will be made for each individual patient at one year after final HBOT session.
  The number of patients who develop recurrent urinary tract infections relative to the total number of patients receiving HBOT and reported as a percentage.
Pre and post treatment symptom survey fro the chronic interstitial cystitis study group. The patient's overall rating of improvement of symptoms (PORIS) will be used. | Three year study period. Determination is made for this endpoint on the date prior to first HBOT and final HBOT session and then by telephone followup at 1, 6, and 12 months following the last HBOT session.
  The PORIS has three questions that address the overall change in CIC/PBS, pain, and urgency after treatment as worse, no better (0% improvement), slightly improved (25%), moderately improved (50%), greatly improved (75%), or symptoms gone (100% improvement). Responders will be defined as those individuals with scores falling into the moderately or greatly improved or no symptoms categories. The number of responders will be reported as a percentage of total number of individuals completing 40 HBOT sessions.
Time of occurrence of recurrent urinary tract infection. | Three year study period. Determination of this endpoint will be made for each individual patient at one year after final HBOT session.
  The time in days at which a recurrent urinary tract infection is occurs will be recorded from the date following final HBOT session and reported as a mean with standard deviation.

CONTACTS AND LOCATIONS:
Overall Officials: Ian R Grover, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Hillcrest Hosptial, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared. Summarized/group data will be shared between sponsor-investigator and Co-PI's at conclusion of patient enrollment. Data will be obtained by prospective collection and analysis.

REFERENCES:
- [Background] Camporesi EM. Side effects of hyperbaric oxygen therapy. Undersea Hyperb Med. 2014 May-Jun;41(3):253-7. PMID 24984321
- [Background] Propert KJ, Mayer RD, Wang Y, Sant GR, Hanno PM, Peters KM, Kusek JW; Interstitial Cystitis Clinical Trials Group. Responsiveness of symptom scales for interstitial cystitis. Urology. 2006 Jan;67(1):55-9. doi: 10.1016/j.urology.2005.07.014. PMID 16413332
- [Result] Plafki C, Peters P, Almeling M, Welslau W, Busch R. Complications and side effects of hyperbaric oxygen therapy. Aviat Space Environ Med. 2000 Feb;71(2):119-24. PMID 10685584